CLINICAL TRIAL: NCT06594796
Title: A Combined Lifestyle Intervention Delivered by Physio/exercise Therapists for Patients with Persistent Low Back Pain and Overweight or Obesity: a Randomized Controlled Trial with Parallel Economic Evaluation
Brief Title: A Combined Lifestyle Intervention Delivered by Physio/exercise Therapists for Patients with Persistent Low Back Pain and Overweight or Obesity
Acronym: Back2Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Willeke Boonstra (Other)
Responsible Party: Sponsor-Investigator, Willeke Boonstra, PhD candidate, VU University of Amsterdam
Organization: VU University of Amsterdam (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL85373.028.23
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Lifestyle Intervention
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Personnel who analyze the data collected from the study are not aware of the treatment applied to any given group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined lifestyle intervention with LBP care (Experimental): A combined lifestyle intervention (GLI) integrated into standard care for LBP according to clinical guidelines of the Dutch physiotherapy (KNGF) and delivered by GLI certified physio/exercise therapists. A GLI aims to increase physical activity, improve diet and sleep, change health behavior, and are effective in reducing weight amongst overweight and obese adults. The intervention is tailored to the patient's lifestyle risk and clinical LBP factors using shared decision-making. Patients define their own treatment goals and remain in charge of the treatment procedures. The intervention has a duration of two years of which the first six months focus on behavioral change, the latter 18 months focus on maintenance of newly set behaviors. Participants are guided using group and individual sessions where evidence-based behavioral change techniques will be employed such as motivational interviewing, self-monitoring and action and coping planning.
  Interventions: Behavioral: Combined lifestyle intervention and LBP care (physiotherapy, exercise therapy)
- Usual care (No Intervention): Usual care as prescribed by the medical specialist. This can vary from a watchful waiting strategy to referral to physiotherapy, exercise therapy, or general practitioner care according to the Dutch physiotherapy (KNGF) and general practice (NHG) guidelines for LBP; e.g. education, exercise therapy and pain medication. It may also involve re-entry to the hospital after failed treatment in primary care.

INTERVENTIONS:
Behavioral: Combined lifestyle intervention and LBP care (physiotherapy, exercise therapy) — One of five recognized combined lifestyle interventions (BeweegKuur, CooL, SSIB, SLIMMER, X-Fittt) integrated with LBP care.
  Arms: Combined lifestyle intervention with LBP care

SUMMARY:
Low back pain (LBP) is the leading cause of disability worldwide and is costly. Lifestyle factors, such as physical inactivity, stress, sleep, excess weight, and an unhealthy diet contribute to the burden of LBP and the associated increasing demand for care. Moreover, approximately 65% of LBP patients who visit the hospital are overweight. This group is considered a complex patient group. Of the LBP patients who visit the hospital, 74% are referred back to primary care as medical specialists cannot offer them high value care. Targeting both lifestyle factors (e.g., physical activity, sleep and stress) and clinical factors related to low back pain (e.g., muscle strength, endurance, mobility) is important in the management of this group of LBP patients to improve important outcomes (e.g., functioning, physical activity) and reduce costs. Addressing lifestyle factors may also offer additional health benefits like decreased risks of diabetes and cardiovascular diseases.

The primary objective of this project is to improve the management of this complex group of LBP patients, that is, patients who are overweight or obese and who are referred back to primary care from the hospital because medical specialists cannot offer them high value care, and to reduce healthcare and societal costs. The primary research question is: 'Is a combined lifestyle intervention, integrated into standard care for LBP, delivered by physio/exercise therapists effective and cost-effective in improving physical functioning and/or physical activity over a 36-month period compared to usual care in overweight or obese LBP patients who are referred back from the hospital to primary care?' It is hypothesized that the combined lifestyle intervention, integrated into standard care for LBP, is both effective and cost-effective in managing LBP in patients who are overweight or obese over a 36-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent (≥3 months) non-specific LBP who are referred back from the hospital to primary care
* Either BMI≥30 OR BMI≥25 with at least one comorbidity (osteoarthritis, sleep apnea, risk factors for cardiovascular diseases or type 2 diabetes)
* Decreased physical functioning (RMDQ ≥4 out of 24)
* Average LBP intensity of ≥3 out of 10 over the past week (NPRS)
* ≥18 years old

Exclusion Criteria:

* Specific LBP (e.g., tumor or fracture)
* Back surgery in the past six months
* Psychiatric diseases that could hinder participation
* Pregnancy or ≤9 months postpartum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Physical activity will be assessed by the activPAL as the average number of daily steps over a period of one week. | Baseline, 6, 24 and 36 months. Primary outcome 36 months.
  The activPAL is a small non-invasive electronic logger designed to quantify free-living daily activities. The activPAL measures physical activity and sedentary behaviour through measuring accelerations and posture of the thigh.
Physical functioning will be measured using the Roland Morris Disability Questionnaire (RMDQ). | Baseline, 6, 12, 24 and 36 months. Primary outcome 36 months.
  The RMDQ is a reliable tool to measure the impact of LBP on physical functioning. It is a 24-item self-report questionnaire about how low back pain affects functional activities. Each question is worth one point, therefore scores can range from 0 (no disability) to 24 (severe disability).

SECONDARY OUTCOMES:
Low back pain levels will be assessed by the Numeric Pain Rating Scale (NPRS) | Baseline, 6, 12, 24 and 36 months
  The NPRS is a 11-point scale consisting of integers from 0 to 10; 0 representing "no pain" and 10 represents "worst possible pain".
Weight and BMI | Baseline, 6, 12, 24 and 36 months
  Weight will be objectively measured via a standardized procedure using the same scale throughout the study. Weight status will be classified using Body Mass Index by dividing body weight (kg) by height (m²).
Sleep quality and duration will be assessed with the Pittsburg Sleep Quality Index (PSQI) | Baseline, 6, 12, 24 and 36 months
  The PSQI consists of 19 items that cover seven dimensions, including subjective sleep quality, sleep duration and latency (time it takes to fall asleep), and the frequency and severity of specific sleep-related complaints in the previous month. Scores from each dimension (range: 0-3) are summed to derive a sleep quality score, higher scores indicate worse sleep quality.
Habitual food intake will be assessed with a Food Frequency Questionnaire (FFQ) | Baseline, 6, 12, 24 and 36 months
  The FFQ is an adapted version of the Dietary Instrument for Nutrition Education. It consists of 20 food items and has a reference period of one month.
A process evaluation will be conducted alongside the RCT with a mixed-method approach. | Baseline, 6 and 24 months
  The process evaluation will study the implementation and mechanism of impact of the intervention. Both participants and physio/exercise therapists will be asked to fill in questionnaires at baseline, 6 and 24 months. A selection of participants will be invited to join a focus group and a selection of physio/exercise therapists will be invited for a semi-structured interview about their experiences during the intervention.
Systemic inflammation (TNF-alpha, hsCRP) | Baseline, 12 and 36 months
  Three times, one vacutainer (7ml blood) will be extracted using venipuncture and serum will be stored at -80 degrees Celcius untill all data has been collected. Serum inflammatory concentrations (TNF-alpha, hsCRP) will be measured using highly sensitive ELLA by an experience laboratory technician. The choice of inflammatory markers may change before analyses due to new insights.
Quality of Life (QALYs) | Baseline, 6, 12, 24 and 36 months
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that measures a participants' health state across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems". The participants' health states will be converted into utility values using the Dutch tariff, after which Quality Adjusted Life Years (QALYs) will be calculated by multiplying the participants spent in a certain health state by the respective utility value (45). In addition, each subject will rate their own perceived health status on a visual analogue scale (VAS) of 0 to 100.
Costs will be measured using a questionnaire based on various iMTA questionnaires. | Baseline, 3, 6, 9, 12, 18, 24, 30 and 36 months
  Costs will be measured from a societal and a healthcare perspective. From the societal perspective, costs will include the cost of the intervention, other healthcare use (i.e., primary, secondary, and medication), informal care, sports memberships and equipment, as well as the cost of productivity losses from paid (i.e. absenteeism and presenteeism) and unpaid work. From the healthcare perspective, only costs accruing to the formal Dutch healthcare sector will be included. Intervention costs will be micro-costed, meaning that detailed data will be collected regarding the number of resources used and their respective unit prices. For this, data will be gathered from questionnaires filled in by participating physio/exercise therapists. Information on all other kinds of resource use will be collected using cost questionnaires. These questionnaires are based on the various iMTA questionnaires but tailored to the specific patient population and intervention under study.
Global perceived effect will be measured using a 7-point scale consisting of integers 1 through 7. | 6, 12, 24 and 36 months
  Each point on the scale indicates a different level of improvement; 1 representing "very much improved", 2 representing "much improved", 3 representing "minimally improved", 4 representing "no change", 5 representing "minimally worse", 6 representing "much worse" and 7 represent "very much worse". Participants will be asked to rate their overall status since the start of the study. The participants' responses to the GPE will be dichotomized into "Recovered" (1 and 2), and "Not Recovered" (3, 4, 5, 6, and 7).

OTHER OUTCOMES:
Pain beliefs will be assessed using the Brief Illness Perception Questionnaire (B-IPQ) | Baseline
  The B-IPQ is a tool used to evaluate cognitive and emotional representations of illness. It is an 8-item questionnaire where each item is rated on a 0-10 scale, with higher scores indicating a more threatening perception of the illness. Total score can be between 0 and 80, higher scores indicate worse illness perception. Cut-off points for the B-IPQ total score as follows: <42 indicating low experienced threat, 42-49 indicating moderate experienced threat, and ≥50 indicating high experienced threat in patients.
Pain self-efficacy will be assessed using the Pain Self-Efficacy Questionnaire (PSEQ) | Baseline
  The PSEQ is developed to assess the confidence people with ongoing pain have in performing activities while in pain. The PSEQ is applicable to all persisting pain presentations. The questionnaire consists of 10 questions scored between 0 (no confidence) and 6 (full confidence). Total score can be between 0 and 60, where a higher score indicates greater levels of confidence in dealing with pain.
Kinesiophobia will be assessed using the Tampa scale for kinesiophobia | Baseline
  The Tampa scale for kinesiophobia is a 17-item questionnaire which are scored between 1 (low fear of movement) and 4 (high fear of movement). Total score can be between 17 and 68. A score ≤37 is interpreted as absence of fear of movement, a score of >37 is interpreted as fear of movement.
Socio-economic status | Baseline
  Education will be considered as a fundamental indicator of socioeconomic status.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyne Scholten-Peeters, PhD, PT, Principal Investigator — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands